CLINICAL TRIAL: NCT06005701
Title: Mallampati Score for Prediction and Prognosis of Postoperative Mortality and Morbidity and Safety Profiles of Patients Undergoing Laparoscopic Cholecystectomy in Qassim Region
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Qassim University (Other)
Responsible Party: Principal Investigator, Mohammed Abaalkhayl, Assistant Professor, Qassim University
Other Study IDs: 23-33-05
Record Dates: First submitted 2023-08-15; First posted 2023-08-22 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Mallampati Score; Difficult Intubation; Patient Satisfaction; Cholestasis; Cholecystitis
Keywords: Mallampati Score; Surgery; Anesthesia
MeSH Terms: conditions — Patient Satisfaction; Cholestasis; Cholecystitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To predict the majority of Mallampati score for the patients in Qassim region who undergoing Laparoscopic Cholecystectomy Surgery.

DETAILED DESCRIPTION:
A preoperative assessment by anaesthetic staff should include the Mallampati Score, as there is a direct correlation between the amount of space in the pharynx and the laryngoscopic view during intubation which has been refined by Cormack and Lehane (1984) Clinical diagnosis one of most important factor indicating the postoperative complications like Mallampati score. As the Mallampati class zero per se is not indicating with any difficulty of airway management unless other airway characteristics indicating to the difficulty. As well as if the epiglottis may be large and overhanging, it's not common with airway difficulty in Mallampati class zero airway.

The Mallampati score idea is to estimate the size of the tongue related to the oral cavity and the displacement of the tongue by the laryngoscope blade was likely to be easy or difficult. It also assessed whether the mouth could be opened adequately to permit intubation

Research objectives To predict the majority of Mallampati score for the patients in Qassim region who undergoing Laparoscopic Cholecystectomy Surgery.

Method:

Observational, Multi hospital, Regional Study

Inclusion Criteria:

1. Age: 20 - 50 years
2. Laparoscopic Cholecystectomy Surgery
3. Body Mass Index (BMI): ≤ 35

Exclusion Criteria:

1. Age Less than 20 years
2. Age More than 50 years
3. Body Mass Index (BMI) > 35

Data management and analysis plan:

All data will be entered and analyzed using SPSS V28© (IBM Corp., Armonk, NY, USA). Categorical variables will have expressed as frequencies and percentages, while continuous variables will have presented as means ± standard deviations (SDs). The chi-squared test will have used to evaluate demographic and health-related characteristics associated with name of the clinic as well as type of service provided to the patient. A p-value of less than 0.05 was considered to be statistically significant

Ethical considerations:

* All investigators completed the Bioethics certificate from The National Committee of Bioethics at King Abdulaziz City for Science and Technology.
* All investigators declare there is no conflict of interest.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 20 - 50 years
2. Laparoscopic Cholecystectomy Surgery
3. Body Mass Index (BMI): ≤ 35

Exclusion Criteria:

1. Age Less than 20 years
2. Age More than 50 years
3. Body Mass Index (BMI) > 35

Ages: 20 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: All patients underwent or planned for Laparoscopic Cholecystectomy
Sampling Method: Probability Sample
Enrollment: 470 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Surveillance | 3 months
  predict the majority of Mallampati score for the patients in Qassim region who undergoing Laparoscopic Cholecystectomy Surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Qassim University Medical City, Buraidah, Al-Qassim Region, Saudi Arabia